CLINICAL TRIAL: NCT03966638
Title: Clinical and Radiological Evaluation of Meniscal Healing After Percutaneous Intra-meniscal
Brief Title: Clinical and Radiological Evaluation of Meniscal Healing After Percutaneous Intra-meniscal Injection of Platelet-rich Plasma (PRP)
Acronym: COMPARE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2019_006
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Meniscus Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving platelet rich plasma: The group is composed of patients receiving an intra-meniscal injection of platelet-rich plasma, under echographic control, for isolated meniscal lesion.
  Interventions: Procedure: Intra-meniscal injection of platelet-rich plasma

INTERVENTIONS:
Procedure: Intra-meniscal injection of platelet-rich plasma — Intra-meniscal injection of platelet-rich plasma under echographic control

SUMMARY:
Meniscal lesions are a common pathology among athletes, and have an impact on the daily or sporting practice of patients. The consequences of surgical treatment are sometimes heavy.

Platelet-rich-plasma (PRP) has been shown to be effective in healing tendon and ligament lesions.

PRP has been injected under ultrasound in tendons or intra-articularly for several years.

This technique of meniscal percutaneous injection of PRP is now carried out for more than 2 years in our hospital, with satisfactory preliminary results, without any complication.

All patients in our study received an intra-meniscal injection of PRP, under echographic control. They were evaluated clinically and by Magnetic Resonance Imaging (MRI) before and at 6 months of the injection.

The aim of the study is to evaluate the efficacy of intra-meniscal injection of PRP on the symptomatology of the patients (pain, sport activities and daily life) at 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* isolated symptomatic meniscal lesion
* lesion confirmed by MRI
* grade II or III lesion touching the peripheral involvement of the middle segment,
* lesion treated by percutaneous intra meniscal PRP's injection
* IKDC score measured before injection and 6 months post-injection

Exclusion Criteria:

* other painful etiology of the knee
* emergency surgical management (luxation, bucket handle) or not (indication validated by the surgeon, meniscectomy or meniscal suture)
* impossibility to perform the procedure (non visible lesion, morphology of the patient, cutaneous infection, coagulation treatment in progress)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with symptomatic non-surgical meniscal injury treated with percutaneous intravenous injection of platelet-rich plasma (PRP)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Variation of International Knee Documentation Committee (IKDC) score | Between 0 and 6 months post injection
  The variation of IKDC score between before injection and 6 months post-injection will be calculated. The IKDC score ranges from 0 to 100 and is interpreted as a measure of function with higher scores representing higher levels of function.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No